CLINICAL TRIAL: NCT00664573
Title: Assessment of Safety and Efficacy of BG9924 in Subjects With RA Who Have Participated in Study 104RA202.
Brief Title: 104RA204 Assessment of the Safety and Efficacy of BG9924 in Rheumatoid Arthritis (RA) Participants
Acronym: RESPOND-EXT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Analysis of data from 104RA202 failed to meet primary endpoint
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 104RA204; 2007-000733-19 (EudraCT Number)
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Safety; Rheumatoid Arthritis; Baminercept alfa; Methotrexate; BG9924; Efficacy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baminercept; Lymphotoxin-beta

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 2 (Experimental): Drug: BG9924 - dose administered as per Biogen-Idec protocol
  Interventions: Biological: Baminercept alfa (BG9924)
- Group 1 (Experimental): Drug: BG9924 - dose administered as per Biogen-Idec protocol
  Interventions: Biological: Baminercept alfa (BG9924)
- Group 3 (Experimental): Drug: BG9924 - dose administered as per Biogen-Idec protocol
  Interventions: Biological: Baminercept alfa (BG9924)
- Group 4 (Experimental): Drug: BG9924 - dose administered as per Biogen-Idec protocol
  Interventions: Biological: Baminercept alfa (BG9924)

INTERVENTIONS:
Biological: Baminercept alfa (BG9924) — dosage administered as per Biogen-Idec protocol
  Other Names: BG9924; Baminercept alfa; LT beta

SUMMARY:
To observe the long-term treatment with BG9924 when administered to participants with RA who previously participated in a Biogen Idec Study.

ELIGIBILITY:
Inclusion Criteria:

* Must be a participant from Study 104RA202 (NCT 00664716)
* Stable dose of Methotrexate for the duration of the study

Exclusion Criteria:

* Participants with a significant change in their medical history from their previous BG9924 study
* Any clinically significant infectious illness or serious local infection

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To Observe The Long-Term treatment with BG9924 When Administered to Participants with RA who Previously Participated in a Biogen Idec Study | Duration of this study is 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (8):
- Coordinating Research Site, San Miguel de Tucumán, Argentina
- Coordinating Research Site, São Paulo, Brazil
- Coordinating Research Site, Budapest, Hungary
- Coordinating Research Site, Cuernavaca, Mexico
- Coordinating Research Site, Torun, Poland
- Coordinating Research Site, Brăila, Romania
- Coordinating Research Site, Moscow, Russia
- Coordinating Research Site, Leeds, Yorkshire, United Kingdom